CLINICAL TRIAL: NCT01632319
Title: Treatment for Excessive Alcohol Use and Depression in Students (TREADS)
Brief Title: Therapy for Undergraduate College Students Who Binge Drink and Are Depressed
Acronym: TREADS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Paola Pedrelli, Director of Dual Diagnoses Studies, Depression Clinical and Research Program, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2008P001357
Record Dates: First submitted 2012-06-28; First posted 2012-07-02 (Estimated); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Depression; Alcohol Abuse
MeSH Terms: conditions — Depression; Alcoholism | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- MI + CBT (Experimental): Motivational Interviewing (MI) and cognitive behavioral therapy (CBT). In this course of therapy students are asked questions about their drinking, receive personalized feedback about it and are taught coping skills for their depressive symptoms.
  Interventions: Behavioral: Combined Motivational Interviewing and Cognitive Behavioral Therapy
- CBT (Active Comparator): Cognitive behavior therapy (CBT)
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Combined Motivational Interviewing and Cognitive Behavioral Therapy — 8 sessions with study clinician, which focus on depressive symptom treatment and alcohol use Both courses teach coping skills for depression (CBT). However, one course focuses only on treatment for depression whereas the other provides also information tailored to the students' level of drinking and experience with regard to alcohol use.
  In one course students are asked questions about their drinking, receive personalized feedback about it and are taught coping skills for their depressive symptoms
  Arms: MI + CBT
Behavioral: Cognitive Behavioral Therapy — Cognitive behavioral therapy is a type of therapy in which students will be taught coping skills for their depressive symptoms but they may or may not talk about alcohol consumption depending on the students' preference.
  Arms: CBT

SUMMARY:
The purpose of this study is to investigate the effectiveness of 2 different therapy courses for undergraduate college students who binge drink and experience depressive symptoms.

DETAILED DESCRIPTION:
After a screening visit (2 ½ hrs) to confirm eligibility for the study, all participants will receive 8 weekly, 1-hour, individual sessions therapy with a counselor. Participants will be randomly assigned, by chance, like the flip of a coin, to the therapy course they will attend. In one of the therapy courses, students are asked questions about their drinking and receive personalized feedback about it, and are taught coping skills for their depressive symptoms. In the second course, students are also taught coping skills for their depressive symptoms but they may or may not talk about alcohol consumption depending on the students' preference. So, both courses teach the same coping skills for depressive symptoms but include different levels of focus on alcohol.

Participants will also complete 2 follow-up visits, at the end of the 8 sessions and then again 4 weeks after completing treatment. These will involve filling out some questionnaires and completing a few neuropsychological tests (these questionnaires and neuropsychological tests will also be completed during the screening visit).

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled in college as an undergraduate student.
* Ages 18-24 years (inclusive).
* Presence of two binge drinking episodes in the past month (defined as consumption of 5 or more drinks in 2 hours for males and 4 for females; NIAAA, 2004).
* BDI-II 12 (12 is often used to indicate the presence of at least mild depressive symptoms) and <30 (indicating severe depression).

Exclusion Criteria:

* Meeting criteria for substance dependence or abuse (any substance) in the past six months (students with alcohol abuse will not be excluded).
* Diagnosis of bulimia, psychosis, or bipolar disorder.
* Having received any psychosocial treatment for depression or substance abuse in the past month.
* Having received CBT for depression and/or alcohol use in the previous 6 months.
* If receiving pharmacological treatment for depression or substance abuse, has not been on a stable dose for at least 4 weeks.
* Discontinued an antidepressant medication less than 1 month ago.
* Meeting criteria for severe depression or posing a serious suicide or homicide risk.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2012-05; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Daily Drinking Questionnaire | 8 weeks
  A measure assessing how much one drinks in a typical week

SECONDARY OUTCOMES:
Beck Depression Inventory | 8 weeks
  A measure assessing symptoms of depression

CONTACTS AND LOCATIONS:
Overall Officials: Paola Pedrelli, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States